CLINICAL TRIAL: NCT04025515
Title: ATORG001 - Molecular Profiling Project
Brief Title: Molecular Profiling Project
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ATORG001
Record Dates: First submitted 2019-06-15; First posted 2019-07-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Oncomine Focus Panel Assay; Molecular profiling; Targeted therapies; Driver oncogene; Next-Generation Sequencing (NGS); PD-L1 Immunohistochemistry (IHC, Dako 22C3); Hotspots; Single Nucleotide Variants (SNVs); Insertions/ Deletions (Indels); Copy Number Variation (CNVs),; Gene Fusions; Formalin-Fixed; Paraffin Embedded (FFPE) extracted DNA and RNA; Ion PGM™ System; Oncomine™ Comprehensive Assay v3
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 unstained FFPE slides of 4 microns per section
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, the investigators plan to undertake comprehensive molecular profiling of "actionable" alterations in lung cancer specimens in order to determine the prevalence of each genetic subtype in the local population.

DETAILED DESCRIPTION:
ATORG is undertaking a comprehensive molecular profiling of "actionable" alterations in lung cancer specimens in order to determine the prevalence of each genetic subtype. These mutations are screened using the Oncomine Focus Assay, where 52 genetic alterations - including hotspots, single nucleotide variants, indels, CNVs, and gene fusions - may be detected in a single workflow. Oncomine™ Comprehensive Assay v3, an NGS assay which tests for 161 unique genes (Appendix IV), will be used in a later stage of the study, allowing for broader coverage of potentially targetable alterations. Both assays have a rapid turnaround time and addresses one of the main challenges of solid tumor testing - the scarcity of tissue material - requiring minimal sample input and thus enabling the use of a wider range of sample quality and types, including small biopsies and fine needle aspirates. However, as the list of therapeutically relevant biomarkers continues to expand over time, broader NGS panels will be used subsequently to incorporate emerging alterations. In addition, relevant baseline clinical characteristics are collated e.g. patient demographics, smoking history, number of lines of therapy, as well as outcomes including access to targeted therapies, immune checkpoint inhibitors and overall survival. Through comprehensive annotation of clinical-pathological-molecular characteristics, this study will provide a means to rationalize the application of diagnostic tests, as well as identify prognostic and predictive factors in the treatment of Asian lung cancers.

ELIGIBILITY:
Inclusion Criteria:

* The availability of sufficient archival tumor tissue specimen (15 slides of 4 microns per section)
* Age ≥ 21 years
* WHO performance status ≤ 2
* Life expectancy of ≥ 12 weeks
* Patients should have adequate organ function for potential consideration into clinical trials (routine blood tests are valid within 14 days before enrollment):

  * Adequate bone marrow function as shown by: ANC ≥ 1.0 x 10^9/L, Platelets ≥ 75 x 10^9/L, Hb ≥ 7.5 g/dL
  * Alanine aminotransferase (ALT) and aspirate aminotransferase (AST) normal range (or ≤3.0 x ULN if liver metastases are present)
* Willing to provide signed informed consent
* Patients whom do not fulfill the above criteria may be discussed on a case-by-case basis with the study team, for potential enrolment

Exclusion Criteria:

- No more than 3 lines of cytotoxic chemotherapy at the time of enrolment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian patients with Non-Small Cell Lung Cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Molecular profiling of lung cancer specimens | After patient meets the eligibility criteria and consent has been taken
  Lung cancer specimens will be collected and profiled at a molecular level to evaluate the molecular epidemiology of NSCLC in Asia

SECONDARY OUTCOMES:
Collection of patient survival status | After molecular profiling has been completed, every few months up to 2 years
Collection of subsequent patient treatment status | After molecular profiling has been completed, every few months up to 2 years
Collection of the clinical outcomes of the subsequent treatments the patients receive | After molecular profiling has been completed, every few months up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tan, BSc, MBBS, MRCP, Principal Investigator — National Cancer Centre, Singapore
Locations (10):
- The Brunei Cancer Centre, Brunei, Brunei
- Hong Kong (2):
  - Hong Kong Integrated Oncology Centre, Hong Kong
  - The Chinese University of Hong Kong, Department of Clinical Oncology, Hong Kong
- Rajiv Ghandhi Cancer Institute and Research Centre, New Delhi, India
- Malaysia (4):
  - Penang Adventist Hospital, George Town
  - Pantai Hospital, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Clinical Oncology Department, Kuala Lumpur
  - Beacon Hospital, Petaling Jaya
- National Cancer Centre Singapore, Singapore, Singapore
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.scri.edu.sg/crn/asian-thoracic-oncology-research-group-atorg/ongoing-research/